CLINICAL TRIAL: NCT00301886
Title: A Phase III Randomized, Multicenter Non-Inferiority Trial Evaluating the Efficacy of Oral Ibandronate Versus Intravenous Zoledronate in the Reduction of Skeletal-Related Events in Patients With Metastatic Breast Cancer
Brief Title: S0308 Zoledronate or Ibandronate in Preventing Bone Problems in Women With Stage IV Breast Cancer That Has Spread to the Bone
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: withdrawn support for study
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000463758; S0308 (Other: SWOG); U10CA037429 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer; Hypercalcemia of Malignancy; Metastatic Cancer; Pain
Keywords: pain; hypercalcemia of malignancy; stage IV breast cancer; bone metastases; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Humoral Hypercalcemia Of Malignancy; Neoplasm Metastasis; Pain | interventions — Ibandronic Acid; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronate (Experimental): zoledronate
  Interventions: Drug: zoledronate; Procedure: quality-of-life assessment
- ibandronate (Experimental): ibandronate
  Interventions: Drug: ibandronate; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: ibandronate
  Other Names: ibandronate sodium
  Arms: ibandronate
Drug: zoledronate
  Other Names: zoledronic acid
  Arms: zoledronate
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Zoledronate and ibandronate may prevent or help relieve bone pain and other symptoms caused by bone metastases. It is not yet known whether zoledronate is more effective than ibandronate in preventing bone problems caused by bone metastases due to breast cancer.

PURPOSE: This randomized phase III trial is studying zoledronate to see how well it works compared to ibandronate in preventing bone problems in women with stage IV breast cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of zoledronate vs ibandronate, in terms of preventing the occurrence of skeletal-related events (SRE) (e.g., fracture, spinal cord compression, radiotherapy or surgery for bone symptoms or events, or hypercalcemia ≥ grade 3), in women with stage IV breast cancer and bone metastases.

Secondary

* Compare the change in patient-reported measures of pain and use of analgesics in patients treated with these drugs.
* Compare the time to first clinically apparent SRE in patients treated with these drugs.
* Compare the toxicity of these drugs.
* Compare the changes in performance status and overall survival of patients treated with these drugs.

OUTLINE: This is a multicenter, randomized study. Patients are stratified according to hormone receptor status (estrogen receptor [ER] and progesterone receptor [PR] negative vs ER and/or PR positive) and current evidence of fracture (vertebral or nonvertebral) or spinal compression (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral ibandronate once daily on days 1-28.
* Arm II: Patients receive zoledronate IV over 15 minutes on day 1. In both arms, treatment repeats every 28 days for up to 18 courses in the absence of unacceptable toxicity.

Quality of life and pain are assessed at baseline, every 3 courses during study treatment, and at the end of study treatment.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 488 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV breast cancer at primary diagnosis or at recurrence

  * Any T, any N, M1
* At least 1 dominant osteolytic or osteoblastic or mixed metastatic lesion outside any prior radiation field

  * Lesion measures ≥ 1.0 cm by x-ray, CT scan, and/or MRI
* Controlled asymptomatic brain metastases allowed
* Controlled bone pain, defined as a physician/health care provider rating of ≤ grade 2 pain-SELECT (Bone) on the NCI CTC for Adverse Events Version 3.0 rating scale, required
* Current evidence of vertebral or nonvertebral fractures or spinal compression due to cancer, as determined by the treating physician, allowed
* No Paget's disease of the bone
* Estrogen receptor (ER) or progesterone receptor (PR) status known

PATIENT CHARACTERISTICS:

* Female patient
* Menopausal status not specified
* Zubrod performance status 0-2
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* Serum calcium < 12 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must be able to receive IV medication and oral medication (i.e., must have physical integrity of the upper gastrointestinal tract)
* No malabsorption syndrome
* No primary hyperparathyroidism
* No known history of aspirin-sensitive asthma
* No other prior malignancy except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I or II cancer currently in complete remission
  * Any other cancer for which the patient has been disease-free for at least 5 years
* No uncontrolled medical illness or infection, including, but not limited to, the following:

  * Unstable angina
  * Recent myocardial infarction
  * Life-threatening cardiac arrhythmia

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bisphosphonates for metastatic bone disease
* More than 28 days since prior aminoglycoside antibiotics
* At least 28 days since prior oral bisphosphonates for osteoporosis
* More than 6 months since prior bisphosphonates used for adjuvant therapy
* Concurrent treatment, including chemotherapy, hormonal therapy, and/or biologic therapy for metastatic breast cancer allowed
* No concurrent participation in another clinical treatment trial for this cancer unless the patient is no longer receiving the intervention and is in the follow-up phase of the other clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Skeletal-related events (SRE)

SECONDARY OUTCOMES:
Change in patient's rating of worst pain as measured by the Brief Pain Inventory
Survival and time to first clinically apparent SRE
Tolerability and toxicity as measured by NCI CTCAE v3.0
Changes in performance status

CONTACTS AND LOCATIONS:
Overall Officials: Saul E. Rivkin, MD, Study Chair — Swedish Cancer Institute at Swedish Medical Center - First Hill Campus; Kathy S. Albain, MD, Study Chair — Loyola University; Dawn Hershman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center